CLINICAL TRIAL: NCT05405569
Title: Influence of Posture and Positioning in Rescuer's Fatigue and Quality of Chest Compressions: a Simulation-based Exploratory Study
Brief Title: Influence of Posture and Positioning in Rescuer's Fatigue and Quality of Chest Compressions
Acronym: QualityCPR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Arcada University of Applied Sciences (Unknown); Centro de Investigação em Tecnologias e Serviços de Saúde (Other); Rede de Investigação em Saúde (Other); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Other Study IDs: QualityCPR
Record Dates: First submitted 2022-05-20; First posted 2022-06-06 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: Cardiopulmonary resuscitation; Chest compressions; Rescuer Fatigue; Quality and performance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Manikin laying on the ground and rescuer kneeled on the floor
  Interventions: Other: CPR Arms Angle 90º; Other: CPR Arms Angle 60º
- Group 2: Manikin laying on a bed at the level of the rescuer knees and rescuer standing on the side of the bed
  Interventions: Other: CPR Arms Angle 90º; Other: CPR Arms Angle 60º
- Group 3: Manikin laying on a higher bed and rescuer standing on a step stool on the side of the bed (the manikin should be at the level of rescuers knees)
  Interventions: Other: CPR Arms Angle 90º; Other: CPR Arms Angle 60º
- Group 4: Manikin laying on a bed and rescuer kneeled on the bed, on the side of the manikin.
  Interventions: Other: CPR Arms Angle 90º; Other: CPR Arms Angle 60º

INTERVENTIONS:
Other: CPR Arms Angle 90º — Within each independent group, a randomized crossover design will be used: half of the group will start with arms position at 90º.
Other: CPR Arms Angle 60º — Within each independent group, a randomized crossover design will be used: half of the group will start with arms position at 60º.

SUMMARY:
Cardiopulmonary resuscitation (CPR) is an emergency maneuver used in a victim who is in cardiac arrest. Early and efficient CPR, with special focus on chest compressions, is a key element to improve patient's survival. The focus for success in resuscitation should not only be the rapid onset of the maneuvers, but also the quality with which they are applied. There are several ways to improve CPR quality, taking training an important role and being relevant for skills acquisition and retention, for both healthcare professionals and laypeople. American Heart Association (AHA) recently recommended the use of technology-enhanced simulators and learning management systems to tailor the training and promote retention. Both training methodologies and support devices are built considering fundamental research, aiming the improvement of patient's outcomes. Based on these scientific developments, guidelines are established focusing on several aspects related to resuscitation, presenting variants of the procedures and considering the profile of the victim. Therefore, studying the quality of CPR and the factors that influence the rescuer's performance is very relevant. The study of fatigue in CPR maneuvers has appeared in the literature mainly after the recent updates to the guidelines. In addition to intrinsic fatigue, there are other extrinsic factors to the CPR maneuver that influence its quality, such as the posture and the position of the rescuer, among others. Most published studies investigate the influence of a single factor in CPR quality, as opposed to the combination of the above-described factors in correlation with rescuer fatigue. We consider this void in literature an opportunity to explore how these factors correlate among them, and how they influence CPR performance and quality. We anticipate that the results from this multi-centre, international project will promote rescuer awareness to specific posture/positioning that influence their fatigue and performance, through the formal development of recommendations to, ultimately, promote high quality CPR. It is expected that this study will provide translational validity, as it is expected to result in changes in current clinical practice.

DETAILED DESCRIPTION:
The aim of this study is to evaluate how positioning and posture of the rescuer promote fatigue and influence the quality of chest compressions. These factors have been selected based on available literature, researchers' experience and feasibility, aiming to answer the research question: in healthcare professionals experienced in CPR, does specific body position and arms angle promote fatigue and influence the quality of chest compressions?

Through this research question we will explore:

1. The influence of positioning during CPR in rescuers fatigue;
2. The influence of the arms angle during CPR in rescuers fatigue; and
3. The correlation between rescuer fatigue during CPR (under specific conditions) and the quality of chest compressions.

It is expected that the conclusions of this research will promote rescuer awareness and behavioral change, leading to better patient outcomes.

Study Design An international multicentric randomized manikin study will be implemented. The protocol development will consider the most recent CONSORT guidelines for randomized clinical trials (RCTs) and the inputs from the experienced research team with formal training in emergency care, simulation-based training, and quantitative research methodology. The protocol will be revised by healthcare professionals, specialized in emergency care and experienced in CPR, from our university hospitals. Formal registration of the protocol will be done to ClinicalTrials.gov. Prior to the study implementation, the study protocol will be submitted for ethical/institutional approval.

Participants will be randomized into 4 independent groups, based on a specific setting/factor:

1. Manikin laying on the ground and rescuer kneeled on the floor;
2. Manikin laying on a bed at the level of the rescuer knees and rescuer standing on the side of the bed;
3. Manikin laying on a higher bed and rescuer standing on a step stool on the side of the bed (the manikin should be at the level of rescuers knees); and
4. Manikin laying on a bed and rescuer kneeled on the bed, on the side of the manikin.

To avoid bias due to the influence of other intrinsic or extrinsic factors, such as height of the rescuer or softness of the mattresses, in all settings, the manikin will be placed at the level of rescuer knees and the mattress will be removed from the bed.

Within each independent group, a randomized crossover design will be used: half of the group will start with arms position at 90º in relation to manikin's chest and the remaining with arms at 60º. Each participant will perform the exercise twice, with a resting period of 10 minutes between exercises. Each exercise consists on 3 minutes of uninterrupted chest compressions. The resting time period between the two arms positions exercises will provide a washout for potential residual effects, such as accumulated fatigue.

Measurements and data collection Participants performance (quality of chest compressions), together with other physical and biological parameters will be evaluated under the above defined conditions. Both single and multi-factor influence will be evaluated to allow studying each factor individually and in combination with others.

Demographic data and baseline physical condition will be collected, using an online questionnaire.

Fatigue will be self-assessed using the Borg Scale, at the end of each 3-minutes exercise. Participants will also self-report fatigue, during the exercise, which will be timed with a chronometer. For heart rate data collection, a standard commercialized heart rate monitor will be used (included in a sports band). Borg Scale was selected as it has a direct relationship with heart rate, allowing a cross-correlation.

Laerdal Resusci Anne QCPR manikin with Laerdal SimPad will be used to assess chest compressions performance parameters (frequency, depth, and recoil). The system will be checked and standardized between participating partners (including mechanical/physical features and software). A standard cardiac arrest clinical scenario will be used. Based on Laerdal software, each CPR session will create a log file that will be used to analyze the performance. The log file will also provide a complete chest compressions waveform to be analyzed using a MATLAB script.

Potentially, the influence of other factors and other observed variables may be explored, if they arise during the study.

Participants selection The sample will be recruited by convenience (nonprobability sample), based on the eligible healthcare professionals (nurses, physicians, paramedics, etc) available to each study partner. Each recruited individual will be submitted to an admission process in order to be considered a participant of the study. Eligibility criteria considers inclusion criteria: (1) Healthcare professionals from 18 to 65 years old; (2) Good general health and physical condition; and (3) Experience in CPR performance, and exclusion criteria: (1) Pregnant women; (2) Exceptional reported physical fatigue and/or muscle pain; and (3) Not being able to read and understand english.

The first step of the admission process is the presentation of the study and the opportunity to provide any clarification needed. An informed consent will be provided and filled voluntarily. Each participant will be assigned with a unique anonymous ID.

The second step is to assess the physical condition by measuring the height, weight, heart rate at rest and physical activity based on the Stanford Brief Activity Survey.

The third step is allowing the participant to use the training manikin for 2 minutes for a self-training session, using automated feedback on the quality of compressions. This will allow each participant to refine performance and to familiarize with the manikin. After this brief training, the participant will fill the sociodemographic questionnaire and the randomization process will be applied (allocation to one of the four settings and selection of the arms position to begin with).

Sample size Sample size was calculated considering 4 independent groups (based on the number of settings) and 2 paired variables (based on the arms position). An ANOVA test, for repeated measures and within-between interactions, was selected to estimate the sample size. Values α = 0.05 and 1-β = 0.80 were considered. The effect size considered was 0.25, based on an estimated medium effect size. An estimate minimum sample size of 48 participants was determined, using G*Power (v3.1.9.7). Ideally, around 60 participants should be recruited anticipating dropouts. Randomization should consider covariates distribution. Based on the established minimum 60 participants, 15 participants should be allocated to each setting.

Statistical analysis Descriptive and inferential statistical analysis will be performed using IBM SPSS Statistics® software, version 28. Sociodemographic data will be used as covariates to assess a homogeneous sample.

Operationalization of the study The project will involve 3 research institutions in 3 countries, envisioning a multi-centre, interdisciplinary approach. This study will provide translational validity, as it may result in new recommendations and changes in current practice.

The data collection will take place in the three involved institutions:

1. Biomedical Simulation Center of the Faculty of Medicine of the University of Porto (Portugal);
2. Human Simulation Center at the Institute for Emergency Medicine and Management in Medicine, Ludwig-Maximilians University Munich (Germany);
3. Patient Safety and Learning Center, ARCADA University of Applied Sciences (Finland).

Each site will be closely monitored by a local expert, following a common detailed protocol and specific equipment, for CPR performance and for data acquisition.

Being a multicentric study, standardization is a key aspect for reliability and validity. The developed protocol was built in close collaboration between partners and several follow up meetings will be planned during the implementation and execution of the study. Site visit to the partner institutions will assure the correct installation of necessary equipment and instruments, and its calibration.

A pilot test will be implemented prior to the full study. This pilot will test the implementation and operationalization of the protocol using a group of elements familiarized with CPR from each partner institution.

ELIGIBILITY:
Inclusion Criteria:

1. Healthcare professionals from 18 to 65 years old;
2. Good general health and physical condition;
3. Experience in CPR performance

Exclusion Criteria:

1. Pregnant women;
2. Exceptional reported physical fatigue and/or muscle pain;
3. Not being able to read and understand english

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample will be recruited by convenience (nonprobability sample), based on the eligible healthcare professionals (nurses, physicians, paramedics, etc) available to each study partner.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in quality of chest compressions | Data collection will be executed continously and synchronized during each CPR session (2 interventions, for 3 minutes each - total 6 minutes) for all participants.
  Laerdal Resusci Anne QCPR manikin with Laerdal SimPad will be used to assess chest compressions performance parameters (frequency, depth, and recoil). A standard cardiac arrest clinical scenario will be used. Based on Laerdal software, each CPR session will create a log file that will be used to analyze the performance. The log file will also provide a complete chest compressions waveform to be analyzed using a MATLAB script. This data will be synchornized with Fatigue data (namely, heart rate data), by starting the recording at the same time in the beginning of each CPR session.
Change in Rescuer's Fatigue | Data collection will be executed continously and synchronized during each CPR session (2 interventions, for 3 minutes each - total 6 minutes) for all participants.
  Fatigue will be self-assessed using the Borg Scale (min. value 6 and maximum value 20, representing "very, very light" and "very, very hard", respectively), at the end of each 3-minutes exercise. Participants will also self-report fatigue, during the exercise, which will be timed with a chronometer. Heart rate data will also be collected and synchronized with chest compressions data - for this, a standard commercialized heart rate monitor will be used (included in a sports band). Borg Scale was selected as it has a direct relationship with heart rate, allowing a cross-correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Sa-Couto, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Faculty of Medicine (FMUP), Porto, Portugal

IPD SHARING:
Plan to Share IPD: No